CLINICAL TRIAL: NCT05511259
Title: Assessing Causality of the Association Between Exercise and Neurocognitive Gains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Responsible Party: Principal Investigator, SH Annabel Chen, PhD, Professor of Psychology, School of Social Sciences, Nanyang Technological University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MOE2019-T2-1-019
Record Dates: First submitted 2022-03-14; First posted 2022-08-22 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2022-08

CONDITIONS: Aging Well
Keywords: healthy aging; older adults; cognition; exercise; neuroplasticity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Intervention group: 3-month community based exercise program (square stepping exercise)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise-Cognition (Experimental): Square Stepping Exercise
  Interventions: Other: exercise
- No exercise (No Intervention): Passive control group

INTERVENTIONS:
Other: exercise — Square stepping exercise
  Arms: Exercise-Cognition

SUMMARY:
Brief Summary: The aim of this project is to examine:

1. The effects of a community based square stepping exercise programme on cognitive and physical functions in older adults.
2. The effects of a community based square stepping exercise programme on neuroplasticity in older adults.
3. The effects of a community based square stepping exercise programme on structural and functional brain changes in older adults.
4. The relationship between exercise-induced changes in neuroplasticity, structural and functional brain activations, and cognitive and physical gains in older adults.

DETAILED DESCRIPTION:
It is well known regular exercise produces both physical and cognitive benefits. Emerging evidence suggests that physical movements or exercise that have concurrent cognitive demands may have more profound effects on cognitive and brain health outcomes. One training program that incorporates these components is the square stepping exercise (SSE). First demonstrated in Japan, this community-based paradigm has already shown to reduce falls risk and presents as a convenient exercise modality for older adults, that can be conducted in a group setting or even the home. The current project aims to examine the efficacy of this SSE community programme in a Singapore context on cognitive and physical health in older adults. This study also aims to quantify the neural correlates underpinning any observed improvements in cognitive and physical function. Specifically, this project will measure indices of neuroplasticity via structural and functional magnetic resonance imaging, transcranial magnetic stimulation, and electroencephalography.

Sample size estimation: n=80 for behavioural primary outcome measures and n=40 subset of larger sample for neuroimaging and neuroplasticity secondary outcome measures [anticipated].

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 55-80
* Sedentary, defined as exercise less than 3 times per week for 30 minutes

Exclusion Criteria:

* Square stepping exercise:
* Medical conditions preventing them from movement and/or exercise
* Psychiatric conditions
* Cognitive impairment of dementia
* Upper and/or lower limb injuries in the past 6 months
* History of falls in the past 6 months
* Current smokers
* Neuroimaging (all the above in addition to the following)
* Patients who have conductive, ferromagnetic, or magnet-sensitive metals implanted in head (e.g., aneurysm clip, stent).
* Implanted medical device: e.g., cardiac implants, cochlear implant, aneurysm clips, cardiac pacemaker etc.
* Non-removable metal braces or retainer (dental fillings ok).
* Permanent tattoos on head.
* Deep brain stimulators.
* Previous brain surgery or injury.
* Patient with epilepsy or any other seizure history, or immediate family history of epilepsy.
* Clinical EEG that was abnormal or where seizure activity had not been ruled out.
* Patients with history of head injury with loss of consciousness are to be investigated about the history if/before being recruited.
* Diagnosis or possibility of neurological disorder (including stroke).
* Psychiatric condition.
* Major or unstable medical condition/surgery.
* Current or suspected pregnancy or lactation.
* Illicit drug use in the last 7 days.
* Alcohol use in the last 12 hours or more than 3 standard drinks in last 24 hours.
* Recent insomnia or severe sleep deprivation.
* Participation in another study involving brain stimulation (e.g., TMS, TDCS) in the past 7 days.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Go-No-Go task change | Baseline (week 0), mid-intervention (week 7 after session 12), post-intervention (week 13 after session 24)
  Error rate: Number of "Go" responses on "No-Go" trials.
Stroop task colour words and colour blocks | Baseline (week 0), mid-intervention (week 7 after session 12), post-intervention (week 13 after session 24)
  Average response time (reaction time) for the correct colour word incongruent trials.
N-Back task change | Baseline (week 0), mid-intervention (week 7 after session 12), post-intervention (week 13 after session 24)
  Number of correct responses (hits)
Trail Making Test ((TMT) change | Baseline (week 0), mid-intervention (week 7 after session 12), post-intervention (week 13 after session 24)
  B:A: Divide the time taken for TMT B by TMT A
Digit Span task change | Baseline (week 0), mid-intervention (week 7 after session 12), post-intervention (week 13 after session 24)
  Maximum accurate span length for Digit Span Forward Maximum accurate span length for Digit Span Reverse
Modified Card Sorting task change | Baseline (week 0), mid-intervention (week 7 after session 12), post-intervention (week 13 after session 24)
  Total number of perseverative errors
Static balance (single leg) change | Baseline (week 0), post-intervention (week 13 after session 24)
  Duration required to perform single leg stance on left and right legs
Temporal gait parameters change | Baseline (week 0), post-intervention (week 13 after session 24)
  11-meter gait test to examine gait speed
Motor learning change | Baseline (week 0), post-intervention (week 13 after session 24)
  Probabilistic Serial Reaction Time Task: learning index, computed using reaction time

SECONDARY OUTCOMES:
Change in cortical thickness | Baseline (week 0), post-intervention (week 13 after session 24)
  T1 and T2 weighted images
Change in grey matter volume | Baseline (week 0), post-intervention (week 13 after session 24)
  T1 and T2 weighted images
Change in structural topography | Baseline (week 0), post-intervention (week 13 after session 24)
  T1 and T2 weighted images
Change in white matter integrity | Baseline (week 0), post-intervention (week 13 after session 24)
  Diffusion Tensor Imaging
Change in white matter connectivity | Baseline (week 0), post-intervention (week 13 after session 24)
  Diffusion Tensor Imaging
Change in functional connectivity | Baseline (week 0), post-intervention (week 13 after session 24)
  Resting state functional magnetic resonance imaging
Brain plasticity changes | Baseline (week 0), post-intervention (week 13 after session 24)
  Changes in transcranial magnetic stimulation (TMS) induced motor evoked potential amplitudes in response to theta-burst stimulation protocol
Brain plasticity changes | Baseline (week 0), post-intervention (week 13 after session 24)
  Changes in transcranial magnetic stimulation (TMS)-evoked potentials recorded from electroencephalography (EEG)
Brain plasticity changes | Baseline (week 0), post-intervention (week 13 after session 24)
  Changes in power spectral density and coherence recorded from electroencephalography (EEG)

OTHER OUTCOMES:
Subjective vitality scale change | Baseline (week 0), post-intervention (week 13 after session 24)
  5-item vitality score (7-point scale, higher score greater wellbeing outcome)
Heart rate variability change | Baseline (week 0), post-intervention (week 13 after session 24)
  Measured through deep breathing protocol with electrocardiography (ECG)
Falls risk change | Baseline (week 0), post-intervention (week 13 after session 24)
  Falls efficiency scale, 16-item and 4-point scale. Lower score equates to more fear of falling and less confident during daily activities.
Social engagement and cohesion | Baseline (week 0), post-intervention (week 13 after session 24)
  Physical Activity Group Environment Questionnaire: 21 items on 9-point scale. Higher scores = more social connection. The community social participation scale will be used as a covariate when analyzing this scale.
Change in mood (related to movement) | Baseline (week 0), post-intervention (week 13 after session 24)
  Anxiety and depression subscale of Movement Specific Reinvestment Scale: 10-item, 6-point for anxiety and depression around movement. Higher scores = more symptoms of anxiety and depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data will be shared after publication and upon request. Request for data needs to justify use of data.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: Request needs to be made to the PI with clear plan for the use of data.